CLINICAL TRIAL: NCT06437353
Title: Sorafenib Combined With Carboplatin/Paclitaxel and Sorafenib Combined With Olaparib as First-line and Maintenance Therapy for Newly Diagnosed High-risk Ovarian Cancer: a Single-arm, Multicenter, Exploratory Clinical Study
Brief Title: Surufatinib Combined With Carboplatin/Paclitaxel and Surufatinib Combined With Olaparib as First-line and Maintenance Therapy for Newly Diagnosed High-risk Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Collaborators: Hutchison Medipharma Limited (Industry)
Responsible Party: Principal Investigator, Bai-Rong Xia, Director of Gynecological Surgery, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024 No. 047
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer
Keywords: Antiangiogenic
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; surufatinib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-line and maintenance therapy regimen (Experimental): First-line chemotherapy regimen:
  * Paclitaxel: 175 mg/m², intravenous infusion, on day 1.
  * Carboplatin: AUC 5, intravenous infusion, on day 1.
  * Surufatinib：250 mg once daily, taken continuously.
  Maintenance Therapy Regimen:
  * Surufatinib: 250 mg once daily, taken continuously.
  * Olaparib: 300 mg twice daily.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — First-line chemotherapy regimen:
  * Paclitaxel: 175 mg/m², intravenous infusion, on day 1.
  * Carboplatin: AUC 5, intravenous infusion, on day 1.
  * Surufatinib：250 mg once daily, taken continuously.
  Maintenance Therapy Regimen:
  * Surufatinib: 250 mg once daily, taken continuously.
  * Olaparib: 300 mg twice daily.
  Other Names: Surufatinib; Carboplatin

SUMMARY:
The goal of this type of clinical trial study is to evaluate the safety and efficacy of Surufatinib combined with Carboplatin/Paclitaxel and Surufatinib combined with Olaparib as first-line and maintenance therapy for newly diagnosed high-risk ovarian cancer

DETAILED DESCRIPTION:
Patients will have tests and exams to see if they are eligible for the clinical trial.

First-line chemotherapy regimen:

Paclitaxel/Carboplatin(repeat every 3 weeks, total of 6 cycles):

* Paclitaxel: 175 mg/m², intravenous infusion, on day 1.
* Carboplatin: AUC 5, intravenous infusion, on day 1.
* For patients aged ≥70 years or those with comorbidities, the paclitaxel dose can be adjusted to 135 mg/m².

Surufatinib(repeat every 3 weeks, total of 5 cycles):

* Surufatinib is not used during the first postoperative cycle.
* Starting from the second postoperative cycle, surufatinib is administered at a dose of 250 mg once daily, taken continuously.

Maintenance Therapy Regimen:

HRD-positive Patients:

* Surufatinib: 250 mg once daily, taken continuously.
* Olaparib: 300 mg twice daily, with doses taken 12 hours apart. Olaparib can be used for a maximum of 2 years.

HRD-negative or HRD Status Unknown Patients:

* Surufatinib: 250 mg once daily, taken continuously.

Treatment continues until the patient experiences disease progression or meets other criteria for discontinuation of the study treatment as specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old (≥18, ≤75)
2. Patients with newly diagnosed FIGO stage III or IV high-grade serous ovarian cancer, high-grade endometrioid carcinoma, primary peritoneal cancer, and/or fallopian tube cancer with high-risk factors for recurrence. High-risk recurrence is defined as follows:

   * FIGO stage III with non-R0 resection;
   * FIGO stage IV;
   * Presence of ascites at initial diagnosis.
3. Patients who have undergone primary debulking surgery (PDS) for ovarian cancer.
4. ECOG performance status score: 0-2.
5. Postoperative administration time ≤12 weeks.
6. Expected survival of at least 3 months.
7. Major organ function within 7 days prior to treatment meets the following criteria:

   * Hemoglobin (HB) ≥90 g/L;
   * Absolute neutrophil count (ANC) ≥1.5×10⁹/L;
   * Platelets (PLT) ≥100×10⁹/L.
8. Biochemical parameters must meet the following standards:

   * Total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN);
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN, or ≤5×ULN if liver metastases are present;
   * Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr) ≥60 ml/min.
9. Women of childbearing potential must use effective contraception.
10. Subjects must voluntarily join the study and sign the informed consent form (ICF).
11. Subjects are expected to have good compliance and the ability to follow up on efficacy and adverse reactions as required by the protocol.

Exclusion Criteria:

1. Previous treatment with anti-angiogenic drugs such as apatinib, sorafenib, anlotinib, bevacizumab, or other anti-angiogenic therapies.
2. Pregnant or breastfeeding women.
3. Patients who have previously participated in other clinical trials that have not yet concluded.
4. Patients with evidence or history of significant bleeding tendencies or events within 3 months before enrollment (bleeding >30 mL, accompanied by hematemesis, melena, or hematochezia), hemoptysis (≥5 mL of fresh blood within 4 weeks), or thromboembolic events (including stroke and/or transient ischemic attack) within 12 months.
5. Patients with uncontrolled hypertension (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg).
6. Patients with grade I or higher myocardial ischemia or infarction, arrhythmias (including QTc ≥480 ms), or ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification).
7. Patients with active or uncontrolled severe infections (≥CTC AE grade 2).
8. Patients with renal failure requiring hemodialysis or peritoneal dialysis.
9. Patients with a history of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases, or those with a history of organ transplantation.
10. Patients with persistent proteinuria (≥++) on two consecutive urine tests, and confirmed 24-hour urine protein >1.0 g.
11. Patients with psychiatric disorders, including epilepsy, dementia, severe depression, mania, etc.
12. Patients with any signs or history of bleeding disorders, regardless of severity; patients who experienced any bleeding or hemorrhagic event ≥CTCAE grade 3 within 4 weeks before enrollment; patients with unhealed wounds, ulcers, or fractures.
13. Patients who had arterial or venous thrombotic events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism, within the past 6 months.
14. Patients with symptomatic brain metastases or those whose symptoms have been controlled for less than 2 months.
15. Patients with a history of substance abuse that cannot be relinquished or those with psychiatric disorders.
16. Patients with difficulty swallowing or known absorption disorders affecting drug intake.
17. Patients allergic to treatment drugs sorafenib or paclitaxel/carboplatin.
18. Any other condition that the researcher deems unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-05-25 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12-month
  Progression-free survival on first-line and maintenance therapy with Surufatinib Combined With Carboplatin/Paclitaxel and Surufatinib Combined With Olaparib

SECONDARY OUTCOMES:
Overall Response Rate (ORR | 3-month
  ORR is defined as the proportion of participants achieving Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST (v.1.1). Per RECIST 1.1, CR is defined as the disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of diameters (SoD) of target lesions
Disease control rate | 3-month
  the percentage of patients with complete response, partial response, and stable disease for more than 4 weeks in which response can be evaluated
Overall survival | 3-years
  the date of enrollment to the date of death from any cause
Adverse event | 3-month
  Adverse medical events in clinical trial subjects treated with Surufatinib Combined With Carboplatin/Paclitaxel and Surufatinib Combined With Olaparib

CONTACTS AND LOCATIONS:
Overall Officials: Bairong Xia, Doctor, Study Chair — Anhui Provincial Cancer Hospital; Wenjing Jiang, Study Director — Anhui Provincial Cancer Hospital
Locations (1):
- Anhui Cancer Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No